CLINICAL TRIAL: NCT00767884
Title: Effect of Panretinal Photocoagulation on Optic Nerve Head Topography and Nerve Fiber Layer Parameters
Brief Title: Effect of Panretinal Photocoagulation on Optic Nerve Head Topography
Acronym: PRP
Status: Terminated | Type: Observational
Why Stopped: Low subject recruitment
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0413-08-EP
Record Dates: First submitted 2008-10-03; First posted 2008-10-07 (Estimated); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Diabetic Retinopathy
Keywords: panretinal photocoagulation; diabetic retinopathy; optic nerve head changes
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the optic nerve head changes consequent to panretinal photocoagulation done for diabetic retinopathy.

DETAILED DESCRIPTION:
Panretinal photocoagulation thermally ablates the retina to effect the regression of the neovascular process seen with diabetic retinopathy.2-6 Photocoagulative damage also damages the nerve fiber layer in the process. Since this should theoretically be associated with loss of nerve fibers it is expected to manifest as changes in optic nerve head cupping. There is no available literature to support this hypothesis. In fact the only available study done of the subject refuted the hypothesis.7 The study had a retrospective design and was done before any of the current technology to evaluate optic nerve head morphology was available.

Patients with concurrent glaucoma and diabetes often undergo panretinal photocoagulation as a part of their diabetes treatment. Optic disc cupping is a standard outcome measure for glaucoma diagnosis and progression. If PRP were to cause increased cupping, this can be a significant confounder in determining glaucoma progression based on optic nerve cupping. The findings of the study will help us determine as to how much cupping can be attributed to the PRP, if any at all.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with proliferative diabetic retinopathy or severe non-proliferative diabetic retinopathy otherwise undergoing panretinal photocoagulation for treatment.

Exclusion Criteria:

* Any patient with uncontrolled glaucoma (IOP above target on any occasion in the preceding 6 months) or other optic neuropathy that may confound the analysis of optic nerve head morphology.
* Patients with media opacities (significant cataract, corneal opacity, vitreous hemorrhage) precluding imaging of the optic nerve.
* No PRP done in the previous 6 months.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ophthalmology Clinic at UNMC
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2008-10-29 (Actual); Primary Completion 2013-10-17 (Actual); Study Completion 2013-10-17 (Actual)

PRIMARY OUTCOMES:
Changes in optic nerve head topography before and after panretinal photocoagulation | 3 years
  Compare changes in optic nerve head topography before and after panretinal photocoagulation (PRP)

CONTACTS AND LOCATIONS:
Overall Officials: Vikas Gulati, MD, Principal Investigator — UNMC
Locations (2):
- United States (2):
  - UNMC Truhlsen Eye Institute, Omaha, Nebraska
  - University of Nebraska Medical Center Eye Clinic, Omaha, Nebraska